CLINICAL TRIAL: NCT00551421
Title: A Phase I/II Trial of Pertuzumab in Combination With Cetuximab and Irinotecan in Previously Treated Metastatic Colorectal Cancer
Brief Title: Pertuzumab and Cetuximab in Treating Patients With Previously Treated Locally Advanced or Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00241; 07-070; U01CA062490 (NIH)
Record Dates: First submitted 2007-10-30; First posted 2007-10-31 (Estimated); Results first posted 2015-02-23 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2014-07

CONDITIONS: Adenocarcinoma of the Colon; Adenocarcinoma of the Rectum; Recurrent Colon Cancer; Recurrent Rectal Cancer; Stage III Colon Cancer; Stage III Rectal Cancer; Stage IV Colon Cancer; Stage IV Rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms | interventions — pertuzumab; 2C4 antibody; Cetuximab; Irinotecan; Immunohistochemistry; In Situ Hybridization, Fluorescence; Gene Expression Profiling; Polymerase Chain Reaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (Experimental): Phase I: Patients receive pertuzumab IV over 30-60 minutes on day 1. Patients also receive cetuximab IV over 60-120 minutes on days 2, 8, and 15 of course 1 and on days 1, 8, and 15 in all subsequent courses. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Phase II: Patients receive treatment as in phase I. Pertuzumab is administered at the recommended phase II dose (determined in phase I).
  Interventions: Biological: pertuzumab; Biological: cetuximab; Drug: irinotecan hydrochloride; Other: immunohistochemistry staining method; Other: fluorescence in situ hybridization; Other: gene expression analysis; Other: mutation analysis; Other: polymerase chain reaction; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: pertuzumab — Given IV
  Other Names: 2C4 antibody; monoclonal antibody 2C4; Perjeta; rhuMAb-2C4
Biological: cetuximab — Given IV
  Other Names: C225; C225 monoclonal antibody; IMC-C225; MOAB C225; monoclonal antibody C225
Drug: irinotecan hydrochloride — Given IV
  Other Names: Campto; Camptosar; CPT-11; irinotecan; U-101440E
Other: immunohistochemistry staining method — Correlative study
  Other Names: immunohistochemistry
Other: fluorescence in situ hybridization — Correlative study
  Other Names: fluorescence in situ hybridization (FISH)
Other: gene expression analysis — Correlative study
Other: mutation analysis — Correlative study
Other: polymerase chain reaction — Correlative study
  Other Names: PCR
Other: laboratory biomarker analysis — Correlative study

SUMMARY:
Monoclonal antibodies, such as pertuzumab and cetuximab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Giving pertuzumab together with cetuximab may kill more tumor cells. This phase I/II trial is studying the side effects and best dose of pertuzumab when given together with cetuximab and to see how well they work in treating patients with previously treated locally advanced or metastatic colorectal cancer

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety, tolerability, and recommended phase II dose of pertuzumab when administered in combination with cetuximab in patients with cetuximab-refractory locally advanced or metastatic colorectal cancer.

II. To evaluate the objective tumor response rate (RR) in patients treated with this regimen.

SECONDARY OBJECTIVES:

I. To evaluate the median progression-free survival (PFS) of patients treated with this regimen.

II. To evaluate the median overall survival (OS) of patients treated with this regimen.

III. To evaluate the RR, PFS, and OS in a subgroup of patients who are EGFR-positive by immunohistochemistry.

IV. To explore the relationship between skin rash and the efficacy outcomes of RR, PFS, and OS in these patients.

V. To explore the relationship between objective tumor response on positron emission tomography (PET) scan after course two and the efficacy outcomes of RR, PFS, and OS in these patients.

VI. To explore the relationship between a variety of laboratory correlates and the efficacy outcomes of RR, PFS, and OS in these patients.

OUTLINE: This is a multicenter, phase I dose-escalation study of pertuzumab followed by a phase II study.

PHASE I: Patients receive pertuzumab IV over 30-60 minutes on day 1. Patients also receive cetuximab IV over 60-120 minutes on days 2, 8, and 15 of course 1 and on days 1, 8, and 15 in all subsequent courses.

Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

PHASE II: Patients receive treatment as in phase I. Pertuzumab is administered at the recommended phase II dose (determined in phase I). Previously collected tumor tissue samples are analyzed for correlative studies. Samples are analyzed for KRAS mutations via polymerase chain reaction and pyrosequencing; EGFR expression via immunohistochemistry and fluorescent in situ hybridization (FISH); HER receptor and ligand gene expression; and circulating tumor cells. Additional blood samples are collected periodically to isolate circulating tumor cells and are analyzed via FISH analysis.

After completion of study treatment, patients are followed at 30 days and then periodically thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a history of colorectal cancer (CRC) treated by surgical resection and who develop radiological or clinical evidence of metastatic disease do not require separate histological or cytological confirmation of metastatic disease unless 1 of the following criteria are met:

  * More than 5 years has elapsed between the primary surgery and the development of metastatic disease
  * The primary cancer was stage I
* Patients must have representative tumor specimens in paraffin blocks or at least 15 unstained slides with an associated pathology report obtained at any time prior to study entry:

  * Cytology specimens are not acceptable replacements
* Patients must have their tumor tissue screened for KRAS mutation status, and be found to have a KRAS wild-type tumor:

  * No KRAS-mutated tumor
* Locally advanced or metastatic disease
* Not curable by surgery or amenable to radiotherapy with curative intent
* Must have received an cetuximab-containing regimen for at least 6 weeks for treatment of metastatic disease
* Documented progression of disease or intolerable toxicity during or within 3 months of receiving this regimen
* Patients who have received an cetuximab-containing regimen as adjuvant therapy for resected stage II or III CRC are eligible provided recurrent disease is documented < 6 months after completion of adjuvant treatment
* Must have received >= 1 prior chemotherapeutic regimen for treatment of metastatic disease with any of the following:

  * Cetuximab
  * Must have resolution of any skin rash related to prior treatment with cetuximab
  * No prior cetuximab which required a dose reduction for toxicity
  * 5-fluorouracil or capecitabine
  * Irinotecan hydrochloride or oxaliplatin
* Measurable disease by CT scan or physical exam
* ECOG performance status (PS) 0-1 (Karnofsky PS 70-100%)
* Life expectancy > 12 weeks
* Absolute neutrophil count >= 1,500/mcL
* Platelet count >= 100,000/mcL
* Leukocytes >= 3,000/mcL
* Hemoglobin >= 9 g/dL (transfusion, erythropoietin, or other approved hematopoietic growth factors allowed)
* Total bilirubin =< 1.5 times upper limit of normal (ULN)
* AST and ALT =< 5 times ULN
* Creatinine normal OR Creatinine clearance >= 60 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception prior to and during study therapy
* Cardiac left ventricular ejection fraction >= 50% OR >= lower limit of normal
* No evidence of left ventricular wall motion abnormalities as measured by ECHO or MUGA scan
* None of the following cardiac conditions:

  * Uncontrolled high blood pressure
  * Unstable angina
  * Symptomatic congestive heart failure
  * Congestive heart failure, cardiac dysfunction, or cardiomyopathy requiring medication treatment
  * Myocardial infarction within the past 6 months
  * Serious uncontrolled cardiac arrhythmia
  * New York Heart Association class III or IV heart disease
* No active or uncontrolled infection
* No predisposing colonic or small bowel disorders in which the symptoms are uncontrolled as indicated by baseline pattern of > 3 loose stools/day (in patients without a colostomy or ileostomy)
* Patients with a colostomy or ileostomy may be eligible at investigator discretion
* No psychiatric illness/social situation that would limit compliance with study requirements
* No other prior or concurrent malignancy, except for adequately treated basal cell or squamous cell skin cancer, in situ carcinoma of the cervix, lobular carcinoma in situ in one breast, or other cancer from which the patient has been disease-free for at least 5 years
* No other medical or psychiatric disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the study results or render the patient at high risk for treatment complications
* No history of allergic reactions, hypersensitivity, or intolerance to cetuximab, and/or compounds of similar chemical or biologic composition to pertuzumab or cetuximab (i.e., other monoclonal antibodies such as bevacizumab) that led to discontinuation of the drug
* Patients able to tolerate subsequent infusions after a reaction are eligible
* At least 4 weeks since prior major surgery (e.g., laparotomy) and recovered (Insertion of a vascular access device is not considered major or minor surgery)
* At least 2 weeks since prior minor surgery and recovered (Insertion of a vascular access device is not considered major or minor surgery)
* At least 4 weeks since prior major radiotherapy (e.g., chest or bone palliative radiotherapy)
* At least 4 weeks since prior bevacizumab
* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin C) and recovered
* No prior agents directed against EGFR and/or HER2
* No more than one prior treatment regimen for metastatic disease; Prior chemotherapy in the adjuvant setting following resection of stage II or III disease allowed provided the regimen did not contain irinotecan hydrochloride and/or an agent directed against EGFR and/or HER2
* No prior doxorubicin or liposomal doxorubicin at doses > 360 mg/m^2; epirubicin at doses > 720 mg/m^2; mitoxantrone at doses > 120 mg/m^2; or idarubicin at doses > 90 mg/m^2
* No prior radiotherapy to > 15% of the bone marrow
* No prior standard adjuvant chemoradiotherapy for rectal cancer
* No phenytoin, phenobarbital, carbamazepine, or any other enzyme-inducing anti-convulsant drugs (EIACDs) for at least 7 days before, during, and for 7 days after the final dose of irinotecan hydrochloride
* Concurrent gabapentin or other non-EIACDs are allowed
* No St. John's wort for at least 14 days before, during, and for 7 days after the final dose of irinotecan hydrochloride
* No concurrent corticosteroids, except for stable doses of prednisone (< 20 mg/day or equivalent), topical or inhaled corticosteroids, or corticosteroids for reasons unrelated to treatment of colorectal cancer
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No concurrent filgrastim (G-CSF) or sargramostim (GM-CSF) for any of the following reasons:

  * To avoid dose reductions or delays
  * Prophylactic treatment
  * Treatment of febrile neutropenia
* No other concurrent HER family-targeted therapy
* No concurrent rifampin
* No concurrent herbal remedies unless initiated prior to study entry
* No other concurrent investigational agents
* No other concurrent anticancer therapy, including cytotoxic chemotherapy, radiotherapy, immunotherapy, hormonal therapy, or biological anticancer therapy
* Histologically or cytologically confirmed adenocarcinoma of the colon or rectum
* Site of the primary lesion must be or have been confirmed endoscopically, radiologically, or surgically to be or have been in the large bowel
* No known brain metastases
* No concurrent fluconazole

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2007-10; Primary Completion 2010-11 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kimmie Ng, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 3 patients were enrolled into the original protocol between 11/07 and 05/08. 1 subject developed Grade 3 diarrhea, all 3 subjects experienced significant skin toxicity. The protocol was therefore amended to recruit cetuximab-refractory mCRC patients only. 14 patients were enrolled in this part of the study between 03/09 and 07/10 at 6 US centers.
Pre-assignment Details: One patient enrolled into the amended part of the protocol withdrew consent prior to receiving any study drug.
Groups:
- Pertuzumab and Cetuximab: Original Protocol, Phase I: Patients receive pertuzumab IV over 30-60 minutes on day 1 of each cycle (loading dose cycle 1 only). Patients also receive cetuximab IV over 60-120 minutes on days 2 (loading dose only), 8, and 15 of cycle 1 and on days 1, 8, and 15 in all subsequent cycles. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Amended Protocol, Phase I: Same as Original Protocol (see above) without a loading dose of Cetuximab (maintenance dose given on cycle 1, day 2 instead).
  Phase II: Patients receive treatment as in phase I. Pertuzumab is administered at the recommended phase II dose (determined in phase I).
  Given IV: irinotecan hydrochloride, pertuzumab, cetuximab
  Correlative Studies: laboratory biomarker analysis, gene expression analysis, fluorescence in situ hybridization, mutation analysis, polymerase chain reaction, immunohistochemistry staining method
Period: Original Protocol, Dose Level 1
Arm/Group | Pertuzumab and Cetuximab
Started | 3
Completed | 3 (1 subject developed Grade 3 diarrhea, all 3 subjects experienced significant skin toxicity.)
Not Completed | 0
Period: Amended Protocol (Cetuximab-refr. mCRC)
Arm/Group | Pertuzumab and Cetuximab
Started | 14
Completed | 13
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- Pertuzumab and Cetuximab: Phase I: Patients receive pertuzumab IV over 30-60 minutes on day 1. Patients also receive cetuximab IV over 60-120 minutes on days 2, 8, and 15 of course 1 and on days 1, 8, and 15 in all subsequent courses. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
Arm/Group | Pertuzumab and Cetuximab
Number analyzed (Participants) | 17
Age, Continuous [Median (Full Range); unit: years] | 60 [46 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Recommended Phase II Dose of Pertuzumab When Administered in Combination With Cetuximab (Phase I)
Description: The regimen was deemed intolerable so there was no recommended phase II dose.
Time Frame: 28 days
Measure: Number
Arm/Group | Pertuzumab and Cetuximab
Number analyzed (Participants) | 14
Value | NA — The regimen was deemed intolerable so there was no recommended phase II dose.

2. Primary Outcome: Objective Tumor Response Rate Defined as the Proportion of Patients With a Best Overall Response of CR or PR, Per RECIST Criteria (Phase II)
Description: Objective tumor response rate defined as the proportion of patients with a best overall response of CR or PR, per RECIST criteria (Phase II).
Time Frame: Best tumor response from time period of start of study treatment to study discontinuation.
Measure: Number; unit: percentage of patients
Groups:
- Arm I: Phase I: Patients receive pertuzumab IV over 30-60 minutes on day 1. Patients also receive cetuximab IV over 60-120 minutes on days 2, 8, and 15 of course 1 and on days 1, 8, and 15 in all subsequent courses. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Phase II: Patients receive treatment as in phase I. Pertuzumab is administered at the recommended phase II dose (determined in phase I).
  pertuzumab: Given IV
  cetuximab: Given IV
  irinotecan hydrochloride: Given IV
  immunohistochemistry staining method: Correlative study
  fluorescence in situ hybridization: Correlative study
  gene expression analysis: Correlative study
  mutation analysis: Correlative study
  polymerase chain reaction: Correlative study
  laboratory biomarker analysis: Correlative study
Arm/Group | Arm I
Number analyzed (Participants) | 7
percentage of patients
  Confirmed Partial Response | 14
  Best Response of Stable Disease | 29
  Best Response of Progressive Disease | 57

3. Secondary Outcome: Progression-free Survival
Description: The duration of time from start of study treatment to time of objective disease progression or death.
Time Frame: The duration of time from start of study treatment to time of objective disease progression or death.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I
Number analyzed (Participants) | 7
months | 2.1 [1.5 to 4.9]

4. Secondary Outcome: Overall Survival
Description: The duration of time from start of study treatment to death from any cause.
Time Frame: The duration of time from start of study treatment to death from any cause.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I
Number analyzed (Participants) | 7
months | 3.7 [1.6 to 7.9]

ADVERSE EVENTS:
Time Frame: Adverse event information was collected between November 2007 and October 2010.
Description: 3 patients were enrolled to Dose Level 1. 1 subject developed gr. 3 diarrhea (hospitalized), and skin toxicity was seen among the 3 subjects. The study was amended and the loading dose of cetuximab was eliminated. We report the adverse event results of the subjects enrolled on the original and the amended protocol.
Groups:
- Pertuzumab and Cetuximab: Original Protocol: Patients received pertuzumab IV over 30-60 minutes on day 1 of each cycle (loading dose on cycle 1, day 1 only). Patients also receive cetuximab IV over 60-120 minutes on days 2 (loading dose), 8, and 15 of cycle 1 and on days 1, 8, and 15 in all subsequent cycles. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Amended Protocol, Phase I: Same as the Original Protocol (see above) except the Cetuximab loading dose was no longer given on cycle 1, day 2 (maintainance dose given).
  Phase II: Patients receive treatment as in phase I. Pertuzumab is administered at the recommended phase II dose (determined in phase I).
  Given IV: pertuzumab, cetuximab, irinotecan hydrochloride
  Corrlateive studies: immunohistochemistry staining method, fluorescence in situ hybridization, gene expression analysis, mutation analysis, polymerase chain reaction, laboratory biomarker analysis
Arm/Group | Pertuzumab and Cetuximab
Serious Adverse Events (participants affected / at risk) | 13/16
Other Adverse Events (participants affected / at risk) | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pertuzumab and Cetuximab (N=16)
cardiac ischemia (Cardiac disorders) | 1
troponin elevation (Cardiac disorders) | 1
insomnia (General disorders) | 1
acneiform rash (Skin and subcutaneous tissue disorders) | 1
dry skin (Skin and subcutaneous tissue disorders) | 1
rash/desquamation (Skin and subcutaneous tissue disorders) | 8
skin pain (Skin and subcutaneous tissue disorders) | 3
small bowel obstruction (Gastrointestinal disorders) | 1
diarrhea (Gastrointestinal disorders) | 4
mucositis or stomatitis (Gastrointestinal disorders) | 5
AST elevation (Metabolism and nutrition disorders) | 1
hyperbilirubinemia (Metabolism and nutrition disorders) | 1
hyperglycemia (Metabolism and nutrition disorders) | 1
hypoalbuminemia (Metabolism and nutrition disorders) | 1
hypokalemia (Metabolism and nutrition disorders) | 1
hypophosphatemia (Metabolism and nutrition disorders) | 1
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
hand-foot reaction (Skin and subcutaneous tissue disorders) | 1
dehydration (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pertuzumab and Cetuximab (N=16)
fatigue (General disorders) | 13
fever without neutropenia (General disorders) | 2
insomnia (General disorders) | 2
rigors/chills (General disorders) | 3
weight loss (General disorders) | 2
weakness (non-neuropathic) (General disorders) | 1
acneiform rash (Skin and subcutaneous tissue disorders) | 4
dry skin (Skin and subcutaneous tissue disorders) | 2
edema of head and neck (Skin and subcutaneous tissue disorders) | 2
edema of limb (Skin and subcutaneous tissue disorders) | 3
edema trunk/genital (Skin and subcutaneous tissue disorders) | 1
erythema multiforme (Skin and subcutaneous tissue disorders) | 3
lymphedema (Skin and subcutaneous tissue disorders) | 1
nail changes (Skin and subcutaneous tissue disorders) | 4
other (Skin and subcutaneous tissue disorders) | 1
pruritis (Skin and subcutaneous tissue disorders) | 7
rash/desquamation (Skin and subcutaneous tissue disorders) | 5
skin (other) (Skin and subcutaneous tissue disorders) | 1
abdominal pain (Gastrointestinal disorders) | 6
anorexia (Gastrointestinal disorders) | 7
constipation (Gastrointestinal disorders) | 1
dehydration (Gastrointestinal disorders) | 2
diarrhea (Gastrointestinal disorders) | 6
distension/bloating (Gastrointestinal disorders) | 1
dyspepsia (Gastrointestinal disorders) | 1
esophagitis (Gastrointestinal disorders) | 1
mucositis or stomatitis (Gastrointestinal disorders) | 5
nausea (Gastrointestinal disorders) | 8
vomiting (Gastrointestinal disorders) | 4
incontinence - urinary (Renal and urinary disorders) | 1
proteinuria (Renal and urinary disorders) | 1
vaginal discharge (Reproductive system and breast disorders) | 1
anemia (Blood and lymphatic system disorders) | 9
leukopenia (Blood and lymphatic system disorders) | 2
lymphopenia (Blood and lymphatic system disorders) | 1
thrombocytopenia (Blood and lymphatic system disorders) | 1
urinary tract (Infections and infestations) | 1
colitis - infectious (Infections and infestations) | 1
ALT elevation (Metabolism and nutrition disorders) | 2
AST elevation (Metabolism and nutrition disorders) | 5
alkaline phosphatase elevation (Metabolism and nutrition disorders) | 6
hepatic (other) (Metabolism and nutrition disorders) | 1
hyperbilirubinemia (Metabolism and nutrition disorders) | 1
hyperglycemia (Metabolism and nutrition disorders) | 6
hyperkalemia (Metabolism and nutrition disorders) | 1
hypoalbuminemia (Metabolism and nutrition disorders) | 7
hypocalcemia (Metabolism and nutrition disorders) | 4
hypokalemia (Metabolism and nutrition disorders) | 4
hypomagnesemia (Metabolism and nutrition disorders) | 7
hyponatremia (Metabolism and nutrition disorders) | 4
hypophosphatemia (Metabolism and nutrition disorders) | 4
INR elevation (Metabolism and nutrition disorders) | 1
PTT prolongation (Metabolism and nutrition disorders) | 1
metabolic/lab (other) (Metabolism and nutrition disorders) | 1
back pain (Musculoskeletal and connective tissue disorders) | 1
neuropathy (sensory) (Nervous system disorders) | 3
eyelid dysfunction (Eye disorders) | 1
blurry vision (Eye disorders) | 1
ocular (other) (Eye disorders) | 2
epistaxis (General disorders) | 3
voice changes/dysarthria (General disorders) | 1
depression (Psychiatric disorders) | 1
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
hemoglobin (Blood and lymphatic system disorders) | 2
neutropenia (Blood and lymphatic system disorders) | 1
neurologic (other) (Nervous system disorders) | 1
gastrointestinal (other) (Gastrointestinal disorders) | 1
infection (other) (Infections and infestations) | 1

LIMITATIONS AND CAVEATS:
Combination intolerable due to overlapping toxicities of diarrhea, rash and mucositis; a unique rash with desquamation seen in most patients across all dose levels. Correlative study inconclusive with too few patients and timepoints with results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less